CLINICAL TRIAL: NCT03776123
Title: Post-marketing Surveillance on the Safety of CabometyxTM in Korean Patients Based on "Guideline for Re-examination of New Drugs"
Brief Title: Post-marketing Surveillance on the Safety of CabometyxTM in Korean Patients
Status: Completed | Type: Observational
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: A-KR-60000-021
Record Dates: First submitted 2018-12-10; First posted 2018-12-14 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Renal Cell Carcinoma; Hepatocellular Carcinoma; Differentiated Thyroid Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell; Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this Post Marketing Surveillance (PMS) is to collect and describe safety and effectiveness profile of Cabometyx™ in real clinical practice setting, according to the approved labelling after the approval of marketing authorization.

ELIGIBILITY:
Inclusion Criteria:

* Patients who meet 'Indications' of label for Cabometyx™ as monotherapy
* Patients who are treated with Cabometyx™ for the first time according to label for Cabometyx™ as monotherapy
* Patients who are aged 18 years or older
* Patients who are willing to provide written consent after being informed of this surveillance

Exclusion Criteria:

* Patients who are contraindicated for Cabometyx™ based on Cabometyx™ label

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients administrated Cabometyx™ at the site (Institutions)
Sampling Method: Non-Probability Sample
Enrollment: 347 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2024-03-26 (Actual); Study Completion 2024-03-26 (Actual)

PRIMARY OUTCOMES:
Number of patients experiencing Adverse Events (AEs)/ Serious Adverse Events (SAEs) after Cabometyx™ administration | From baseline until 21 days after the last dose of Cabometyx (up to approximately 52 weeks)
Proportion of patients who had AEs/SAE after Cabometyx™ administration | From baseline until 21 days after the last dose of Cabometyx (up to approximately 52 weeks)
Number of AEs/SAEs after Cabometyx™ administration | From baseline until 21 days after the last dose of Cabometyx (up to approximately 52 weeks)

SECONDARY OUTCOMES:
Objective response rate | From baseline until 21 days after the last dose of Cabometyx (up to approximately 52 weeks)
Progression Free Survival | From baseline until 21 days after the last dose of Cabometyx (up to approximately 52 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (47):
- South Korea (47):
  - Korea University Ansan Hospital, Ansan
  - Hallym University Sacred Heart Hospital, Anyang
  - DONG-A University Hospital (Site A), Busan
  - DONG-A University Hospital (Site B), Busan
  - Kyungpook National University Chilgok Hospital, Daegu
  - Daegu Catholic University Medical Center, Daegu
  - Keimyung University Dongsan Hospital (Site A), Daegu
  - Keimyung University Dongsan Hospital (Site B), Daegu
  - The Catholic University of Korea, Daejeon ST.Mary's Hospital, Daejeon
  - Chungnam National University Hospital, Daejeon
  - Daejeon Eulji Medical center, Eulji University, Daejeon
  - Konyang University Hospital, Daejeon
  - The Catholic University of Korea, Uijeongbu ST. Mary's Hospital (site A), Gyeonggi-do
  - The Catholic University of Korea, Uijeongbu ST. Mary's Hospital (Site B), Gyeonggi-do
  - Chonnam National University Hwasun Hospital, Hwasun
  - Wonkwang University Hospital, Iksan
  - The Catholic University of Korea, St. Mary's Hospital, Incheon
  - Gachon University Gil Medical Center, Incheon
  - Inha University Hospital, Incheon
  - Chungbuk National University Hospital, Jungbuk
  - Inje University Busan Paik Hospital, Pusan
  - Inje University Haeundae Paik Hospital, Pusan
  - Pusan National University Hospital (Site A), Pusan
  - Pusan National University Hospital (Site B), Pusan
  - Kosin University Gospel Hospital (Site A), Pusan
  - Kosin University Gospel Hospital (Site B), Pusan
  - CHA Bundang Medical Center, CHA University, Seongnam
  - Inje University Sanggye Paik Hospital (Site A), Seoul
  - Inje University Sanggye Paik Hospital (Site B), Seoul
  - Korea University Anam Hospital (Site A), Seoul
  - Korea University Anam Hospital (Site B), Seoul
  - Severance Hospital, Yonsei University (Site A), Seoul
  - Severance Hospital, Yonsei University (Site B), Seoul
  - Hanyang University Seoul Hospital, Seoul
  - Gangdong Kyung Hee University Hospital, Seoul
  - Asan Medical Center (Site A), Seoul
  - Asan Medical Center (Site B), Seoul
  - Gangnam Severance Hospital, Yonsei University Health System, Seoul
  - Samsung medical center (Site B), Seoul
  - Samsung Medical Center (Site C), Seoul
  - Samsung Medical Center (Site D), Seoul
  - Samsung Medical Centre (Site A), Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
  - Chung-Ang University Hospital, Seoul
  - The Catholic University of Korea, Yeouido St. Mary's Hospital, Seoul
  - The Catholic University of Korea, St. Vincent's Hospital, Suwon
  - Ulsan University Hospital, Ulsan

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, annotated case report form, statistical analysis plan, and dataset specifications.
  Patient level data will be anonymized and study documents will be redacted to protect the privacy of study participants.
  Any requests should be submitted to www.vivli.org for assessment by an independent scientific review board.
Time Frame: Where applicable, data from eligible studies are available 6 months after the studied medicine and indication have been approved in the US and EU or after the primary manuscript describing the results has been accepted for publication, whichever is later.
Access Criteria: Further details on Ipsen's sharing criteria, eligible studies and process for sharing are available here (https://vivli.org/members/ourmembers/).
URL: https://vivli.org/members/ourmembers/